CLINICAL TRIAL: NCT02271971
Title: Effect of Vitamin D Supplementation on Metabolic Parameters of Patients With Moderate to Severe Psoriasis
Brief Title: Effect of Vitamin D Supplementation on Metabolic Parameters of Patients With Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-412
Record Dates: First submitted 2014-10-19; First posted 2014-10-22 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Psoriasis; Metabolic Syndrome; Vitamin D Deficiency
Keywords: Psoriasis; Vitamin D; Metabolic syndrome; Insulin resistance; Cholesterol; Methotrexate; Dyslipidemia; PASI; Psoriasis Area Severity Index
MeSH Terms: conditions — Psoriasis; Metabolic Syndrome; Vitamin D Deficiency; Insulin Resistance; Dyslipidemias | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 supplementation (Experimental): Subjects in the experimental arm will receive a daily 5.000 IU vitamin D3 capsule during 6 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Subjects in the placebo arm will receive a daily placebo capsule during 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — A daily 5.000 IU vitamin D3 capsule during 6 weeks.
  Other Names: Cholecalciferol
  Arms: Vitamin D3 supplementation
Dietary Supplement: Placebo — A daily placebo capsule during 6 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether supplementation with oral vitamin D (cholecalciferol) improves metabolic parameters in patients with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe psoriasis.
* Being treated with methotrexate with stable doses for al least 1 month.

Exclusion Criteria:

* Phototherapy within the past 2 months.
* History of psoriatic arthritis, rheumatoid arthritis, type 1 diabetes mellitus or inflammatory bowel disease.
* Use of vitamin d supplements or fish oil supplements in the past 2 months.
* Use of hypolipidemic drugs, hypoglycemic drugs, glucose sensitizers, oral corticosteroids, orlistat, cholestyramine, phenobarbital or phenytoin within the past 2 months.
* Pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Total Cholesterol Levels | Baseline and 6 weeks

SECONDARY OUTCOMES:
Change in Fasting Glucose Levels | Baseline and 6 weeks
Change in HOMA Index | Baseline and 6 weeks
Change in Glycated Hemoglobin Levels | Baseline and 6 weeks
Change in Low-Density Lipoprotein Levels | Baseline and 6 weeks
Change in High-Density Lipoprotein Levels | Baseline and 6 weeks
Change in Triglycerides Levels | Baseline and 6 weeks
Change in C-Reactive Protein Levels | Baseline and 6 weeks
Change in Vitamin D Levels | Baseline and 6 weeks
Change in PASI (Psoriasis Area Severity Index) | Baseline and 6 weeks

OTHER OUTCOMES:
Number of Participants with Adverse Events | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Niklitschek, MD, Principal Investigator — School of Medicine, Pontificia Universidad Católica de Chile; Ninoska Porras, MD, Principal Investigator — School of Medicine, Pontificia Universidad Católica de Chile; Hernán Correa, MD, Study Director — School of Medicine, Pontificia Universidad Católica de Chile; Félix Fich, MD, Study Director — School of Medicine, Pontificia Universidad Católica de Chile; Isidora Harz, MD, Study Director — School of Medicine, Pontificia Universidad Católica de Chile; Arturo Borzutzky, MD, Study Director — School of Medicine, Pontificia Universidad Católica de Chile; Luis Villarroel, MD, Study Director — School of Medicine, Pontificia Universidad Católica de Chile; William Romero, MD, Study Director — School of Medicine, Pontificia Universidad Católica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile